CLINICAL TRIAL: NCT02014038
Title: Ultrarunners Longitudinal TRAcking Study (ULTRA)
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: University of California, Davis (Other)
Responsible Party: Principal Investigator, Lorinda S Chung, Assistant Professor of Medicine (Immunology and Rheumatology), Stanford University
Other Study IDs: 21271
Record Dates: First submitted 2013-12-06; First posted 2013-12-17 (Estimated); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Arthritis; Osteoporosis; Injuries
Keywords: Ultrarunners; ultramarathon runners; ULTRA; Physical activity; Health Risks; sedentary; moderately active
MeSH Terms: conditions — Arthritis; Osteoporosis; Wounds and Injuries; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Health status information and physical activity level will be collected longitudinally on a large group of individuals who are ultramarathon runners at the time of enrollment to determine if very high levels of physical activity alter health risks compared with sedentary or moderately active lifestyles.

DETAILED DESCRIPTION:
The intent of this research is to longitudinally study the health of individuals who have run at least one ultramarathon (50K distance or greater) prior to enrollment.Longitudinal data will be collected through periodic (every 1-2 years) survey completion by enrolled subjects over the course of up to 20 years. All surveys will be collected through a secure web-based system used by Stanford University Qualtrics). Minor formatting adjustments will be required when placing into the on-line questionnaire format.

We anticipate that the follow-up surveys will be adjusted prior to use, so they will be submitted to the Institutional Review board as addendum or in continuing review. As indicated elsewhere, subjects will be recruited through an email exchange (referred to as the "Ultralist"), various ultramarathon-related web sites and blogs, and ultramarathon-related magazines. Initial recruitment will continue for up to 12 months or until we have reached our desired sample size. Recruitment material (attached) will include a link to the initial survey. For follow-up surveys, subjects will initially be sent an email (using the address they have provided with the initial survey) that contains a link to the survey and request that they complete the survey. Attempt to contact non-responders will be, in this order, through a second email, phone call, letter to their home, email to identified surrogate, phone call to identified surrogate, and letter to identified surrogate. Publicly available death records will be examined for cases where follow-up cannot be achieved.

ELIGIBILITY:
Inclusion Criteria:Healthy adults, able to provide consent, able to do survey online, must have completed one ULTRA marathon prior to participating in this study.

Exclusion Criteria:Not meeting the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult healthy volunteers who have completed at least one ULTRA marathon (50K distance or greater) prior to enrollment in the study.
Sampling Method: Non-Probability Sample
Enrollment: 2452 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Compare baseline demographic and health (number of lost work days, frequency of various medical conditions, change in BMI with aging) characteristics of ultramarathon runners with published data for less active populations. | Initailly at 12 months from start of enrollment and every one to two years over the next 20 years.
  1. Compare baseline demographic (education level, marital status, amount of TV watching) and health (number of lost work days, frequency of various medical conditions, change in BMI with aging) characteristics of ultramarathon runners with published data for less active populations.
  2. Compare characteristics of those developing various medical conditions over the course of the longitudinal study with those not developing those conditions.
  3. Compare the longitudinal risk of developing various medical conditions between ultramarathon runners and those with sedentary or moderately active lifestyles. Knowledge gained from this work will help define if there is an upper limit in activity level for which health benefits are achieved.

CONTACTS AND LOCATIONS:
Overall Officials: Eswar Krishnan, MD, Principal Investigator — Stanford University; Martin Hoffman, MD, Principal Investigator — University of California, Davis
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States